CLINICAL TRIAL: NCT00296608
Title: Preoperative Radiotherapy With or Without Concurrent Chemotherapy (5-Fluorouracil and Leucovorin) in T3-4 Rectal Cancers - Randomized Trial
Brief Title: Radiation Therapy With or Without Chemotherapy Before Surgery in Treating Patients With Stage II or Stage III Rectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000466625; FFCD-9203; EU-20600
Record Dates: First submitted 2006-02-24; First posted 2006-02-27 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-05

CONDITIONS: Colorectal Cancer
Keywords: stage II rectal cancer; stage III rectal cancer; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Fluorouracil; Leucovorin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiotherapy (Active Comparator): RT was delivered with photons from a linear accelerator with an energy level of 8MVor above.
  Interventions: Procedure: conventional surgery; Radiation: radiation therapy
- Chemotherapy and radiotherapy (Experimental): The first CT cycle was administered from days 1 to 5 of the RT treatment. LV 20 mg/m2/d was delivered intravenously immediately before administration of FU. FU 350 mg/m2/d was delivered during 20 minutes in 100 mL of saline infusion, 1 hour before RT. The second cycle was administered from days 29 to 33 of the RT treatment using the same schedule.
  Interventions: Drug: fluorouracil; Drug: leucovorin calcium; Procedure: conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Drug: fluorouracil
  Arms: Chemotherapy and radiotherapy
Drug: leucovorin calcium
  Arms: Chemotherapy and radiotherapy
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as fluorouracil and leucovorin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving radiation therapy and chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving chemotherapy after surgery may kill any tumor cells that remain after surgery. It is not yet known whether radiation therapy is more effective with or without chemotherapy when given before surgery for rectal cancer.

PURPOSE: This randomized phase III trial is studying radiation therapy given together with fluorouracil and leucovorin to see how well they work compared to giving radiation therapy alone before surgery in treating patients with stage II or stage III rectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the recurrence-free and overall survival of patients with resectable stage II or III adenocarcinoma of the rectum treated with neoadjuvant radiotherapy with or without concurrent chemotherapy comprising fluorouracil and leucovorin calcium followed by surgery and adjuvant fluorouracil and leucovorin calcium.

OUTLINE: This is a randomized, controlled, multicenter study. Patients are stratified according to participating center, gender, location of the tumor relative to the anal margin (0-5 cm vs > 5 cm), and tumor stage (T3 vs T4). Patients are randomized to 1 of 2 treatment arms.

* Neoadjuvant therapy: Patients are randomized to 1 of 2 neoadjuvant therapy arms.

  * Arm I: Patients receive leucovorin calcium IV and fluorouracil IV over 15 minutes on days 1-5. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients also undergo concurrent radiotherapy 5 days a week for 5 weeks.
  * Arm II: Patients undergo radiotherapy as in arm I.
* Surgery: In both arms, patients undergo surgical resection within 3-10 weeks after completing neoadjuvant therapy.
* Adjuvant therapy: Within 3-10 weeks after surgery, all patients receive adjuvant chemotherapy comprising leucovorin calcium IV and fluorouracil IV over 15 minutes on days 1-5. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 6 months for at least 5 years.

PROJECTED ACCRUAL: A total of 762 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the rectum meeting 1 of the following stage criteria:

  * Stage T3, N0-2, M0 disease meeting 1 of the following criteria:

    * Invasive disease in entire circumference (circular tumor)
    * Tumor fixed laterally or posteriorly to pelvic structures
    * Tumor adherent to the prostate and/or seminal vesicles
    * Tumor infiltration into the vaginal-rectal septum
    * Tumor classified as uT3 by rectal endoscopy
  * Stage T4, N0-2, M0 disease meeting 1 of the following criteria:

    * Clinical or radiologic evidence of pelvic organ extension (vagina, prostate, seminal vesicles, or bladder)
    * Tumor extension to the anal canal or sphincter
    * Tumor classified as uT4 by rectal endoscopy
* Tumor accessible by digital rectal exam
* Resectable disease
* No distant metastases

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Creatinine < 1.36 mg/dL
* Granulocyte count > 2,000/mm^3
* Platelet count > 130,000/mm^3
* No progressive ischemic cardiomyopathy
* No acute or chronic obstruction unless treated with diversion colostomy
* No chronic inflammation of the ileum and/or colon
* No other prior or concurrent malignancy except basal cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy, radiotherapy, or surgery for this cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 762 (Actual)
Dates: Start 1993-04; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Gerard, MD, Study Chair — Centre Antoine Lacassagne

REFERENCES:
- [Background] Bonnetain F, Bosset JF, Gerard JP, Calais G, Conroy T, Mineur L, Bouche O, Maingon P, Chapet O, Radosevic-Jelic L, Methy N, Collette L. What is the clinical benefit of preoperative chemoradiotherapy with 5FU/leucovorin for T3-4 rectal cancer in a pooled analysis of EORTC 22921 and FFCD 9203 trials: surrogacy in question? Eur J Cancer. 2012 Aug;48(12):1781-90. doi: 10.1016/j.ejca.2012.03.016. Epub 2012 Apr 14. PMID 22507892
- [Background] Bonnetain F, Bosset J, Gerard J, et al.: An analysis of preoperative chemoradiotherapy with 5FU/leucovorin for T3-4 rectal cancer on survival in a pooled analysis of EORTC 22921 and FFCD 9203 trials: surrogacy in question? [Abstract] J Clin Oncol 29 (Suppl 15): A-3506, 2011.
- [Result] Methy N, Bedenne L, Conroy T, Bouche O, Chapet O, Ducreux M, Gerard JP, Bonnetain F. Surrogate end points for overall survival and local control in neoadjuvant rectal cancer trials: statistical evaluation based on the FFCD 9203 trial. Ann Oncol. 2010 Mar;21(3):518-524. doi: 10.1093/annonc/mdp340. Epub 2009 Sep 16. PMID 19759186
- [Result] Methy N, Bedenne L, Gerard J, et al.: Surrogate endpoints in neoadjuvant rectal cancer trials: statistical evaluation using data from the FFCD 9203 trial. [Abstract] American Society of Clinical Oncology 2008 Gastrointestinal Cancers Symposium, 25-27 January 2008, Orlando, FL. A-466, 2008.
- [Result] Gerard JP, Conroy T, Bonnetain F, Bouche O, Chapet O, Closon-Dejardin MT, Untereiner M, Leduc B, Francois E, Maurel J, Seitz JF, Buecher B, Mackiewicz R, Ducreux M, Bedenne L. Preoperative radiotherapy with or without concurrent fluorouracil and leucovorin in T3-4 rectal cancers: results of FFCD 9203. J Clin Oncol. 2006 Oct 1;24(28):4620-5. doi: 10.1200/JCO.2006.06.7629. PMID 17008704
- [Result] Gerard J, Romestaing P, Bonnetain F, et al.: Preoperative chemotherapy (CT-RT) improves local control in T3-4 rectal cancers: results of the FFCD 9203 randomized trial. [Abstract] Int J Radiat Oncol Biol Phys 63 (2 Suppl 1): A-4, S2, 2005.